CLINICAL TRIAL: NCT06047015
Title: Immune Response to Irreversible Electroporation (NanoKnife ®) and a Checkpoint Inhibitor With or Without CpG Oligodeoxynucleotides for the Treatment of Stage IV Colorectal Cancer
Brief Title: Irreversible Electroporation (NanoKnife ®) and Immunotherapy for the Treatment of Stage IV Colorectal Cancer
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Saskatchewan (Other)
Responsible Party: Principal Investigator, Mike Moser, Associate Professor of Surgery, University of Saskatchewan
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IREIMMU
Record Dates: First submitted 2023-02-21; First posted 2023-09-21 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Liver Metastasis Colon Cancer
MeSH Terms: interventions — Electroporation; CPG-oligonucleotide

STUDY DESIGN:
Intervention Model Description: This will be a pilot study examining 6 patients treated with IRE and checkpoint inhibitor (first 6, non-randomized) and 6 patients treated with IRE and checkpoint inhibitor and CpG
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- IRE plus Checkpoint Inhibitor (Experimental): Nivolumab: Patients will receive 240 mg nivolumab (dissolved in 250 mL NaCl 0.9%) administered intravenously over 30 minutes. The first dose will take place one or two days before the IRE treatment. The second and third doses will be given 2 and 4 weeks post-IRE. Bloodwork will be done just prior to each treatment.
  IRE is performed in the CT scanner. Patients will receive a general anesthetic, and an ultrasound will be performed to locate the designated metastasis. Ultrasound-guided electrode placement (3 or 4 depending on cancer size, shape, and location) will be performed by interventional radiologist Dr. Chris Wall and the IRE device will be activated and used as per the technique of Martin et al.
  Interventions: Combination Product: IRE plus checkpoint inhibitor
- IRE plus Checkpoint Inhibitor plus CpG Oligodeoxynucleotides (CpG-ODN) (Experimental): Patients will receive 240 mg nivolumab as above and also receive 8 mg of CpG-ODN dissolved in 1 mL normal saline administered peritumorally just before the IRE treatment. Three or four electrodes will be placed using a combination of ultrasound and CT guidance in preparation for treatment. Then using the electrodes as landmarks, injection of ¼ or 1/3 cc of the CpG-ODN solution will be performed near each of the 3 or 4 electrodes to achieve a peritumoral administration of the drug.
  IRE is performed in the CT scanner. Patients will receive a general anesthetic and an ultrasound will be performed to locate the designated metastasis. Ultrasound-guided electrode placement (3 or 4 depending on cancer size, shape, and location) will be performed by interventional radiologist Dr. Chris Wall and the IRE device will be activated and used as per the technique of Martin et al.
  Interventions: Combination Product: IRE plus Checkpoint Inhibitor plus CpG-ODN

INTERVENTIONS:
Combination Product: IRE plus checkpoint inhibitor — Nivolumab: Patients will receive 240 mg nivolumab (dissolved in 250 mL NaCl 0.9%) administered intravenously over 30 minutes. The first dose will take place one or two days before the IRE treatment. The second and third doses will be given 2 and 4 weeks post-IRE. Bloodwork will be done just prior to each treatment.
  Arms: IRE plus Checkpoint Inhibitor
Combination Product: IRE plus Checkpoint Inhibitor plus CpG-ODN — Patients will receive 240 mg nivolumab as above and also receive 8 mg of CpG-ODN dissolved in 1 mL normal saline administered peritumorally just before the IRE treatment. Three or four electrodes will be placed using a combination of ultrasound and CT guidance in preparation for treatment. Then using the electrodes as landmarks, injection of ¼ or 1/3 cc of the CpG solution will be performed near each of the 3 or 4 electrodes to achieve a peritumoral administration of the drug.
  IRE is performed in the CT scanner. Patients will receive a general anesthetic and an ultrasound will be performed to locate the designated metastasis. Ultrasound-guided electrode placement (3 or 4 depending on cancer size, shape, and location) will be performed by interventional radiologist Dr. Chris Wall and the IRE device will be activated and used as per the technique of Martin et al.
  Arms: IRE plus Checkpoint Inhibitor plus CpG Oligodeoxynucleotides (CpG-ODN)

SUMMARY:
The goal of this pilot clinical trial is to learn about the combination of immune boosting drugs and irreversible electroporation (IRE) in patients with colon cancer that has spread to the liver (metastasis). The main questions it aims to answer are:

1. to document the rate of complications associated with combining IRE with immune boosting drugs.
2. After one liver metastasis is treated with IRE and immune boosting drugs, what is the change in the size of the non-IRE-treated liver metastases?
3. What is the immune response (measured in a blood sample) when IRE is combined with one or two types of immune boosting drugs?

DETAILED DESCRIPTION:
Single-centre pilot study of the use of IRE for the treatment of 12 patients with unresectable colorectal liver metastases to assess feasibility and gain preliminary data to inform the design of a larger study.

ELIGIBILITY:
Inclusion Criteria:

1. Biopsy-proven colorectal liver metastases with at least one measuring < 3.5 cm in diameter and accessible to percutaneous IRE such that a complete ablation of the lesion is possible.
2. Prior resection of the colorectal cancer primary.
3. The imaging has been reviewed in multi-disciplinary Rounds and the colorectal liver metastases have been deemed unresectable.
4. Patient has undergone chemotherapy and has not converted to resectable disease.
5. Radiologic evidence of stable disease for at least two months on systemic therapy for colorectal cancer (may have had prior partial response or disease progression)
6. Microsattelite instability (MSI)-stable or mismatch-proficient tumors
7. Patient has HLA phenotype of Human Leukocyte Antigen (HLA) A1 or HLA A2.
8. Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

1. Size of the metastasis being treated with IRE > 3.2 cm or < 2 cm.
2. Size of any non-IRE-treated liver metastasis > 4 cm
3. Pregnancy
4. Major comorbid disease
5. Active autoimmune disease
6. Bone or brain or peritoneal metastases.
7. MSI High disease
8. Patients with cardiac arrhythmia other than rate controlled atrial fibrillation.
9. Metal implant that cannot be removed within 10 cm of the area to be treated.
10. Peritoneal disease.
11. Poor performance status
12. Cirrhosis

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2025-07 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Complications | 30 days
  Complications (Clavien-Dindo classification of complications) at 30 days. The Clavien-Dindo Classification of Complications involves assigning a numbered classification to each complication, from 1-5, with 1 being a complication without need for any intervention required to 5 which is death of the patient. (a higher number indicates a higher severity). This is a validated measure in use for over 25 years.
Complications | 90 days
  Complications (Clavien-Dindo classification of complications) at 90 days. The Clavien-Dindo Classification of Complications involves assigning a numbered classification to each complication, from 1-5, with 1 being a complication without need for any intervention required to 5 which is death of the patient. (a higher number indicates a higher severity). This is a validated measure in use for over 25 years.
Abscopal effect: percent change in non-treated colorectal liver metastasis. | 3 months from the time of IRE
  Two radiologists (one diagnostic and the other interventional) will examine the scans of all patients. They will select a colorectal metastasis from the scan just before the intervention that is between 2-3.2 cm in maximal diameter, accessible to percutaneous ablation, and treatable according to the interventional radiologist's opinion. Another metastasis, with a maximal diameter of less than 4 cm, will be selected to monitor for the abscopal effect (reduction in size of a colorectal liver metastasis that was not treated with IRE).
  After 3 months, the radiologists will review the imaging again. They will assess the treatment mass area for any contrast uptake indicating incomplete ablation. The second metastasis will be measured in the same dimensions as before treatment. The difference in maximal diameter of the second metastasis will be calculated as (diameter before IRE - diameter after IRE) / diameter before IRE and expressed as a percentage.

SECONDARY OUTCOMES:
Tumor-specific immune response: distribution on flow-cytometry plot | Day 8
  Distribution of Carcinoembryonic (CEA)-specific CD8+ T cells, CD4+ T cells, type-1 and 2 macrophages (M1 and M2), regulatory T (Treg) cells on the flow-cytometry plot.
Tumor-specific immune response: serum cytokine concentrations | Day 8
  Interleukin(IL)-2, Interferon (IFN)-α, IFN-γ, IL-10 and Transforming Growth Factor (TGF)-β.
Tumor-specific immune response: distribution on flow-cytometry plot. | Day 14
  Distribution of Carcinoembryonic (CEA)-specific CD8+ T cells, CD4+ T cells, type-1 and 2 macrophages (M1 and M2), regulatory T (Treg) cells on the flow-cytometry plot.
Tumor-specific immune response: serum cytokin concentrations | Day 14
  Interleukin(IL)-2, Interferon (IFN)-α, IFN-γ, IL-10 and Transforming Growth Factor (TGF)-β.
Tumor-specific immune response: distribution on flow-cytometry plot. | Day 30
  Distribution of Carcinoembryonic (CEA)-specific CD8+ T cells, CD4+ T cells, type-1 and 2
Tumor-specific immune response | Day 30
  Interleukin(IL)-2, Interferon (IFN)-α, IFN-γ, IL-10 and Transforming Growth Factor (TGF)-β.
Progression-free survival | 1 year
  Progression-free survival will be determined based on the CT scan conducted after one year. To prove the absence of progression, there should be no contrast uptake in the area that was treated with IRE one year prior, AND the maximal diameter of the second lesion (not treated with IRE) should have increased by less than 10%.
Progression-free survival | 2 years
  Progression-free survival will be determined based on the CT scan conducted after two years. To prove the absence of progression, there should be no contrast uptake in the area that was treated with IRE two years prior, AND the maximal diameter of the second lesion (not treated with IRE) should have increased by less than 10%
Quality of life questionnaire | baseline
  Quality of life using FACT-G (Functional Assessment of Cancer Therapy-General) questionnaire, a 27-item questionnaire, each item to be rated 1-5. The scores are totalled and total scores range from 0-108, with higher scores indicating a higher quality of life.
Quality of life questionnaire | 12 weeks
  Quality of life using FACT-G (Functional Assessment of Cancer Therapy-General) questionnaire, a 27-item questionnaire, each item to be rated 1-5. The scores are totalled and total scores range from 0-108, with higher scores indicating a higher quality of life.
Quality of life questionnaire | 1 year
  Quality of life using FACT-G (Functional Assessment of Cancer Therapy-General) questionnaire, a 27-item questionnaire, each item to be rated 1-5. The scores are totalled and total scores range from 0-108, with higher scores indicating a higher quality of life.

IPD SHARING:
Plan to Share IPD: No